CLINICAL TRIAL: NCT01221688
Title: Evaluation of Sentinel Lymph Node Detection After Neoadjuvant Chemotherapy for Large Operable Breast Cancer
Brief Title: Sentinel Lymph Node Detection After Neoadjuvant Chemotherapy for Large Operable Breast Cancer
Acronym: GANEA2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BRD 09/9-G
Record Dates: First submitted 2010-10-11; First posted 2010-10-15 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer
Keywords: Breast cancer; neoadjuvant chemotherapy; False negative rate; Axillary lymph node dissection; Sentinel lymph node
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Early breast cancer patients treated with neo-adjuvant chemotherapy (NAC) were included. Before NAC, patients with cytologically proven node involvement were allocated into the pN1 group, other patient were allocated into the cN0 group. After NAC, pN1 group patients underwent sentinel lymph node (SLN) and axillary lymph node dissection (ALND); cN0 group patients underwent SLN and ALND only in case of mapping failure or SLN involvement.
Oversight: Data Monitoring Committee: No

ARMS (2):
- group 2 (cN0) (Other): Patients without proven axillary involved nodes will undergo SLN biopsy and a complete axillary level I-II lymphadenectomy only in the case of detection failure or involved SLN and a SLN biopsy alone in the others cases. Patients of this last group will be followed 5 years in order to evaluate the risk of axillary relapse without lymphadenectomy.
  Interventions: Procedure: Axillar Sentinel lymph node biopsy
- group 1 (pN+) (Experimental): group 1 : patients with proven involved axillary nodes will undergo SLN biopsy and complete level I-II axillary lymphadenectomy.
  Interventions: Procedure: SLNB and complete level I-II axillary lymphadenectomy

INTERVENTIONS:
Procedure: Axillar Sentinel lymph node biopsy — Group 2 : Patients without proven axillary involved nodes will undergo SLNB and a complete axillary level I-II lymphadenectomy only in the case of detection failure or involved SLN and a SLNB alone in the others cases. Patients of this last group will be followed 5 years in order to evaluate the risk of axillary relapse without lymphadenectomy.
  Arms: group 2 (cN0)
Procedure: SLNB and complete level I-II axillary lymphadenectomy — group 1 : patients with proven involved axillary nodes will undergo SLNB and complete level I-II axillary lymphadenectomy.
  Arms: group 1 (pN+)

SUMMARY:
Neoadjuvant chemotherapy (NAC) is frequently proposed to patients with large tumours that can be operated in order to increase the chances of breast conservation. After NAC, patients are operated with systematic axillary lymph node dissection (ALND), although more than half of these patients do not have lymph node involvement. These results lead us to consider the indication of the sentinel lymph node (SLN) technique after NAC in order to avoid unnecessary ALND in patients whose SLN is free of involvement.

We need to validate the SLN technique after NAC in patients who have proven lymph node involvement prior to NAC.

GANEA2 is a new trial based on patient treated for a large breast tumor with proven axillary involved nodes. Patients enrolled in this trial will have first an axillary sonography with fine needle punction in case of suspected nodes before NAC. This primary evaluation allow to determine two groups of patients : group 1 (pN+) : patients with proven involved axillary nodes and group 2, patients without proven axillary involved nodes (cN0). Patients of group 1, will undergo SLNB and complete level I-II axillary lymphadenectomy. Patients of group 2 will undergo SLNB and a complete axillary level I-II lymphadenectomy only in the case of detection failure or involved SLN and a SLNB alone in the others cases. Patients of this last group will be followed 5 years in order to evaluate the risk of axillary relapse without lymphadenectomy.

ELIGIBILITY:
Inclusion Criteria:

* T2-T3 operable infiltrating breast carcinoma
* No allergy to Patent Blue
* Pre-operative diagnosis of unifocal infiltrating breast carcinoma.
* Patient planned to be treated by NAC.
* Informed consent.
* Surgery available 4 to 6 weeks after the last chemotherapy course (radical or conservative surgery)

Exclusion Criteria:

* pT4d (inflammatory breast cancer)
* Locally advanced or metastatic breast cancer
* Any previous chemotherapy of contra-lateral breast cancer.
* Breast cancer local relapse
* Previous surgical removal of breast Cancer.
* Inadequate biopsy for pathological analysis.
* Dementia or altered mental disorder
* Pregnant woman or breast feeding or without efficacious contraceptive method.
* Contra-indication to NAC NAC interrupted due to progressive disease.
* Neoadjuvant radiotherapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 958 (Actual)
Dates: Start 2010-07-12 (Actual); Primary Completion 2014-10-27 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
false-negative (FN) rate for the Sentinel Lymph Node Detection | after surgery
  Ratio of the number of FN cases to the total number of patients with at least one lymph node involved, sentinel or not.
  a FN case was defined as a patient with a successful mapping, SLN(s) without any metastasis, and a metastasis in at least one node from the ALND

SECONDARY OUTCOMES:
Detection rate | after surgery
  Percentage of patients with SLN detected and isolated intraoperatively
Sataloff score on breast tumour | after surgery
  The Sataloff classification assesses the response of the NAC on the breast tissue.
  TA: total or almost total therapeutic effect. TB: therapeutic effect > 50%. TC: < 50% therapeutic effect but obvious effect. TD: no therapeutic effect
Sataloff score on lymph nodes | after surgery
  The Sataloff classification assesses the response of the NAC on the lymph nodes NA: clear therapeutic effect, no metastases. NB: no therapeutic effect, no metastases. NC: aspects of therapeutic effect, but presence of metastases. ND: no therapeutic effect, viable metastases.
Homolateral axillary recurrence rate | 5 years post surgery
  Recurrence observed groupe 2 patients (cN0) whitout ALND

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc CLASSE, MD, Principal Investigator — INSTITUT DE CANCEROLOGIE DE L'OUEST
Locations (18):
- France (18):
  - CHU, Angers
  - Institut de Cancerologie de L'Ouest, Angers
  - Institut Bergonié, Bordeaux
  - CHU, Brest
  - Centre Jean Perrin, Clermont-Ferrand
  - CH, La Roche-sur-Yon
  - Centre Oscar Lambret, Lille
  - Centre Léon Berard, Lyon
  - Institut Paoli Calmette, Marseille
  - INSTITUT DE CANCEROLOGIE DE MONTPELLIER Val d'aurelle, Montpellier
  - Institut de Cancérlogie de Lorraine, Nancy
  - Institut Curie, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Lariboisière, Paris
  - HEGP, Paris
  - Institut Curie, Saint-Cloud
  - Institut de cancérologie de l'Ouest, Saint-Herblain
  - ICANS, Strasbourg